CLINICAL TRIAL: NCT06472635
Title: A Retrospective, Multicenter, Single-arm Real-world Study on a New Adjuvant Chemotherapy Combined With Immune Inhibitors for Resectable Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: a Neo-adjuvant Chemotherapy Immunotherapy in Resectable ESCC Study
Acronym: ANACIIRE-1
Status: Active, not recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhengliang.Tu, Director of General Thoracic Surgery Department / Chief Doctor, Zhejiang University
Other Study IDs: IIT20230408B-R2
Record Dates: First submitted 2024-06-16; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: The Neoadjuvant Treatment for Resectable Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research Purpose 1: To evaluate the therapeutic efficacy and safety of neoadjuvant immunotherapy combined with chemotherapy in the treatment of resectable locally advanced esophageal squamous cell carcinoma (ESCC) in the real-world setting.

Research Purpose 2: To analyze the influencing factors of the therapeutic effect of neoadjuvant immunotherapy combined with chemotherapy in the treatment of resectable locally advanced esophageal squamous cell carcinoma (ESCC) in the real-world setting.

Research Purpose 3: To understand the treatment patterns of neoadjuvant immunotherapy combined with chemotherapy in the treatment of resectable locally advanced ESCC in the

DETAILED DESCRIPTION:
Research Purpose 1: To evaluate the therapeutic efficacy and safety of neoadjuvant immunotherapy combined with chemotherapy in the treatment of resectable locally advanced esophageal squamous cell carcinoma (ESCC) in the real-world setting.

Research Purpose 2: To analyze the influencing factors of the therapeutic effect of neoadjuvant immunotherapy combined with chemotherapy in the treatment of resectable locally advanced esophageal squamous cell carcinoma (ESCC) in the real-world setting.

Research Purpose 3: To understand the treatment patterns of neoadjuvant immunotherapy combined with chemotherapy in the treatment of resectable locally advanced ESCC in the

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years (including 18 years old); ECOG 0 or 1; Patients with esophageal squamous cell carcinoma judged to be resectable (including initially non-resectable) by the researcher Received esophageal radical surgery and neoadjuvant immune chemotherapy before surgery Clinical staging belongs to: T1b-4NanyM0;

Exclusion Criteria:

Patients without complete medical information; Received other anti-tumor treatment before surgery; Received radiotherapy treatment; Judged by the researcher, have other conditions unsuitable for participating in this clinical study.

Hide hide Contacts/Locations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal Squamous Cell Carcinoma (ESCC), with a follow-up cutoff date of March 2024, is expected to take 6 months for data cleaning and analysis, and the data collection and analysis are anticipated to be completed in September 2024.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | 12 months
  pCR is defined as the ratio of residual viable tumor cells being 0 in the primary tumor and sampled lymph nodes.

SECONDARY OUTCOMES:
Resection Rate | 12 months
  R0 resection refers to the complete removal of the tumor, with negative microscopic margins, indicating no residual tumor; no cancer cells are found on the cutting line under pathological examination.

OTHER OUTCOMES:
ORR | 12 months
  Defined as the proportion of patients achieving complete response (CR) or partial response (PR) among all patients, with efficacy evaluation based on the RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China